CLINICAL TRIAL: NCT05108597
Title: Effect of Rectal Misoprostol in Reducing Intra-operative Blood Loss During Myomectomy A Randomized Control Trial
Brief Title: Effect of Rectal Misoprostol in Reducing Intra-operative Blood Loss During Myomectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Salma Nisar, Resident OBGYN, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 25102021
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Blood Loss, Surgical; Uterine Myoma
MeSH Terms: conditions — Blood Loss, Surgical; Myofibroma | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: There will be a single trained person who calculated the intra-operative blood loss and was blinded to the randomization of the patients and the use of medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol (Study Group) (Experimental): In study group, 400ug misoprostol will be administered through rectal route, 1 hour before surgery.
  Interventions: Drug: Misoprostol
- No drug (No Intervention): In control group no dose will be administered

INTERVENTIONS:
Drug: Misoprostol — 400ug misoprostol will be administered through rectal route, 1 hour before surgery to assess its effect on intra-operative blood loss during myomectomy
  Other Names: Prosotec
  Arms: Misoprostol (Study Group)

SUMMARY:
A total of 200 women for elective abdominal myomectomy were randomly allocated into two groups.

100 women in experimental group were administered 400ug Misoprostol (2 tablets of Prosotec®) through the rectal route prior to surgery and 100 were in control group, in which no drug was administered.

DETAILED DESCRIPTION:
After getting approval from hospital's ethical committee, patients eligible for the study were recruited in the study according to the selection criteria. Before surgery, after taking informed written consent, patient's detailed history including demographics, parity & BMI was recorded. Uterine size was assessed by bimanual pelvic examination. Patients undergoing myomectomy were randomly divided into 2 groups using lottery method. In experimental group Misoprostol 400ug was administered per rectally prior to surgery. In control group, no drug was administered.

The surgical procedural elements, the surgeon or surgeons performing the procedure and the use of antibiotics as well as anesthetic agents was standardized to remove any bias. Intraoperative blood loss was recorded by a single trained doctor and calculated using visual scale for the abdominal sponges and chest swabs/gauzes used during surgery and blood collected in suction bottle.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status class I-II
2. Intramural or subserosal fibroids - diagnosed on ultrasound
3. Candidates for elective abdominal myomectomy

Exclusion Criteria:

1. Pre-operative Hemoglobin < 10 g/dl
2. Patient who received Danazol or GnRH analogues before surgery
3. No other systemic or metabolic disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | During the surgical procedure
  Intraoperative blood loss will be recorded by a trained doctor and calculated using visual scale for the abdominal sponges and chest swabs/gauzes used during surgery and blood collected in suction bottle.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Nisar, Principal Investigator — Resident OBGYN
Locations (1):
- PEMH, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Overall results will be shared only.